CLINICAL TRIAL: NCT06148597
Title: Effects of M-TAPA Block on Postoperative Pulmonary Functions in Laparoscopic Bariatric Surgery: A Randomized Controlled Study
Brief Title: Effects of M-TAPA Block on Pulmonary Functions
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Çağdaş Baytar, Principal Investigator, Zonguldak Bulent Ecevit University
Other Study IDs: 2023/04-4
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Functions; Pain Management; Obesity, Morbid
Keywords: obesity; pain management; pulmonary functions; respiratory function test
MeSH Terms: conditions — Agnosia; Obesity, Morbid; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group M-TAPA
  Interventions: Procedure: Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA)
- Group Control

INTERVENTIONS:
Procedure: Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) — application local anesthetic between internal oblique and transversus abdominis muscle at the level of 10th costal cartilage
  Groups: Group M-TAPA

SUMMARY:
Adequate postoperative analgesia is difficult to achieve in patients undergoing laparoscopic sleeve gastrectomy (LSG). Epidural anesthesia is technically difficult due to subcutaneous fat, which increases the risk of serious complications. Moreover, patients in this condition often have comorbidities that require anticoagulation therapy. Although ultrasound-guided Transversus Abdominis Plane (TAP) block may be useful, it is still controversial.

Recently, modified thoracoabdominal nerve block via perichondrial approach (M-TAPA) has been reported as a new and promising technique that provides effective analgesia in the anterior and lateral thoracoabdominal wall.

The most common reason for hospitalization after laparoscopic surgery is pain after nausea and vomiting. In addition, superficial and tachypneic breathing resulting from the patient's inability to breathe deeply with pain causes closure of small airways and increase in intrapulmonary shunts, resulting in hypoxia. Postoperative pain management is important not only to prevent pain but also to reduce pulmonary complications that may occur due to changes in lung function and to reduce mortality and morbidity by controlling the stress response.

In this study, The investigators investigated the effect of modified thoracoabdominal nerve block via perichondrial approach (M-TAPA) on pulmonary function in patients undergoing laparoscopic bariatric surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years old

  * ASA I-II-III risk group
  * Patients whose approval was obtained through an informed consent form
  * Will undergo laparoscopic bariatric surgery
  * Patients who will cooperate for the PFT test

Exclusion Criteria:

* <18 years and >65 years

  * ASA ≥ IV
  * 50% below the expected value in SFT
  * Known diaphragmatic paralysis
  * Having had a myocardial infarction within 1 month
  * Dementia or confusion
  * Lack of cooperation
  * Those with respiratory disease
  * Congestive heart failure
  * Unstable hypertension
  * Had thoracoabdominal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 who will undergo ASA I-III laparoscopic bariatric surgery
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
FEV1/FVC ratio | during the procedure
  Pulmonary function

SECONDARY OUTCOMES:
Numerical Rating Scale | during the procedure
  pain assessment tool (minimum: 0, maximum: 10)
opioid consumption | 24 hours after surgery
  need of opioid postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No